CLINICAL TRIAL: NCT06343207
Title: Percussive Therapy Reduced EMG Activity During Calf Raise in Limbs With and Without Chronic Ankle Instability: A Randomized Controlled Trial
Brief Title: Percussive Therapy Reduced EMG Activity During Calf Raise in Limbs With and Without Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Lukáš Michal, MSc. Lukas Michal, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 249637
Record Dates: First submitted 2024-03-21; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Ankle Injuries
Keywords: surface electromyography; ankle injury; lower limb injury
MeSH Terms: conditions — Ankle Injuries; Leg Injuries

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CAI PT (Experimental): Chronic ankle instability patient + percussive therapy intervention
  Interventions: Device: Percussive massage gun therapy
- CAI NOPT (No Intervention): Chronic ankle instability patient + NO percussive therapy intervention (control)
- CON PT (Experimental): Healthy subjects + percussive therapy intervention
  Interventions: Device: Percussive massage gun therapy
- CON NOPT (No Intervention): Healthy subjects + NO percussive therapy intervention

INTERVENTIONS:
Device: Percussive massage gun therapy — Between pre and post-test, there was a one and half minute period during which each participant were in a prone position on a medical examination bed. The experimental PT groups received a 30-second triceps surae massage on each limb, while the control group maintained the same prone position without massage. The massage gun was set to 2100bpm and 1 bar of surface pressure was indicated by the device. The massage gun movement was performed according to the manufactu'er's instructions.
  Other Names: TheraGun
  Arms: CAI PT; CON PT

SUMMARY:
To examine the acute effect of percussive therapy on peak calf muscle activation during standing heel raise in subjects with and without chronic ankle instability (CAI).

DETAILED DESCRIPTION:
Total of 42 subjects in mean age of 23.5 ± 2.5 years participated in this research. From the original of 44 subjects, we had to discard 2 subjects (not finishing the measurement and extremely outlier data). The group was divided into 2 specific subcategories as follows - 21 patients with diagnosed CAI (CAI group; respectively) and the 21 of control group patients (HEALTHY group; respectively), including people who have never injured ankles, nor the ligaments and muscles group surrounding the ankle complex. The information and categorization based on the injury history to specific groups was performed by verbal questioning. The criteria for the CAI group were having had at least two ankle luxation or ankle distortions in the last 2 years as reported by a physician. The HEALTHY group was without this diagnosis. All the individuals involved in the testing underwent a medical examination by a sports physician at least once in a period of one year before testing. Subjects of both genders in both groups were then randomly divided (balanced ratio between male and female participants was kept) into 2 subgroups based on applied PT or not as follows: CAI YES (n=10), CAI NO (n=11), HEALTHY YES (n=10), HEALTHY NO (n=11). The probands were informed about the research process, which they also confirmed by signing an informed consent form according to Declaration of Helsinki. The master thesis research was approved by the ethical committee of Faculty of Physical Education and Sport, Charles University.

Data collection of Total Travelled Way (TTW) of Centre of Pressure (COP) during static postural stability tests was performed by pressure platform FootScan (RS Scan International, Belgium). Pressure sensors located in the platform sense load at frequencies up to 500 Hz. In particular, the parameter of Total Travelled Way of COP in mm (TTW) was evaluated and analyzed the postural stability tests consisted of two bilateral and one unilateral test.

First bilateral test was Close Stand with Open Eyes (OE) in duration of 30 s. Subject was asked to stand on pressure platform as close as possible without touching the feet, ankles, or knees between dominant, and nondominant lower limb. Subject was asked to relax, free both arms besides the body and to stand as stable as possible in duration 30 s, while maximally concentrating on the sticker black point, centered, and located 1,5 m in front wall in the height of the eye level (individually set up). Second test was Close Stand with closed Eyes in duration of 30 s. Besides the same body and posture position, the subject was asked to close both eyes during 30 s stand performance. Third test was unilateral stand on one lower limb, also called Flamingo test in duration of 30 s. Subject was asked to gently bend non-supportive lower limb into the air, approximately to 45° knee flexion. Eyes was open during this test. This test was performed for dominant (FLDOM) and nondominant (FLNON) lower limb separately. Dominance of the lower limb was examined and marked by verbal questioning of lateral preference of lower limb. During flamingo tests, subjects were able to choose which lower limb will be tested first. This was followed by 4 trials of Heel Rise test, which the FS recorded for 6s each. Subject was in close stand (arms free and relaxed beside the body) and by the tester command performed controlled heel rise to maximal available and comfortable height in tempo of 2 s concentric phase, 1 second stay in transfer position, and 2 s eccentric phase. Results of TTW in mm during each test were evaluated by FootScan software and assigned to individual subjects' results sheet in MS Excel (Microsoft, USA).

Data collection of calve muscle activity during static and dynamic postural stability tests was performed by surface electromyography (sEMG) by Trigno Sensors (Delsys Inc., Natick, USA) attached to the m. gastrocnemius vastus lateralis bilaterally by experienced practitioner of the laboratory. After subjects' explanation and agreement, the place of sensor application was cleaned, shaved, and again cleaned with medical cleaning cloth (Medipal, Alcohol Wipes), consequently, the sEMG sensor was attached to measurement place by original adhesive stickers from Delsys manufacturer. sEMG activity was recorded simultaneously in all tests. Sample rate of recorded signal was set at 2048 Hz with a 16-bit A/D resolution. Bandwidth of sEMG sensors was high-passed (4th-order Buterworth) at 20±5 hz and low-passed (4th-order Buterworth) at 450±5 hz for further analysis. Further sEMG data analysis was performed by EMGworks Analysis software (Delsys Inc., Natick, USA). Recorded and filtered sEMG data underwent rectification to absolute values and enveloped by window length (root mean squared; RMS) of 200 ms. For EMG activation normalization of DOM and NON lower limb individually, peak RMS muscle activity during flamingo tests (for dominant and nondominant individually) was used and applied to represent the mean RMS in percentages of sEMG activity during each test and each lower limb (%RMSmax). Using unilateral standing on one leg (Flamingo) was preferred before maximal voluntary contraction (MVC) tests of calf muscles, in order to avoid excessive muscle excitation before and during static tests and before PT application.

There was a pause (1:30min) between the 1st and 2nd measurements, during which the experimental group received triceps surae massage for 30s each. The percussive massage gun was set at 2100bpm and the pressure on the surface was 1 bar showed by the device, as indicated by the manufacturer.n During the massage the sEMG sensor were replaced for the easier access to the whole muscle group. After that it was attached to the same place as it was before. Putting it to the same spot was simplified by the fact there were visible pressure marks. The control group laid down to the same position as the experimental one and stayed like that for the same amount of time (1:30min). Afterwards they were tested once again.

ELIGIBILITY:
Inclusion Criteria:

CAI group - at least two ankle luxation or ankle distortions in the last 2 years as reported by a physician.

Healthy group - healthy

Exclusion Criteria:

* paraplegia,
* women in advanced stages of pregnancy
* feverish or acute inflammatory diseases within 7 days before the measurement
* current or healed rupture of m. gastrocnemius, m. soleus, tendo calcaneus
* purulent, fungal diseases, burns, scalds, varices

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Percussive Therapy Reduced EMG Activity During Calf Raise in Limbs With and Without Chronic Ankle Instability. | 1 week
  Recorded and filtered sEMG data by Trigno Sensors (Delsys Inc., Natick, USA) underwent rectification to absolute values and enveloped by window length (root mean squared; RMS) of 200 ms (Farfan et al., 2010). For EMG activation normalization of DOM and NON lower limb individually, peak RMS muscle activity during flamingo tests (for dominant and nondominant individually) was used and applied to represent the mean RMS in percentages of sEMG activity during each test and each lower limb (%RMSmax).

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Michal, MSc., Principal Investigator — Department of Pathophysiology, Charles University, Second Faculty of Medicine
Locations (1):
- Faculty of physical education and sport, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No